CLINICAL TRIAL: NCT03736148
Title: Acute Effects of Manual vs Instrument-assisted Single Cervical Manipulation on Electromyographic Activity and Sympathetic Nervous System
Brief Title: Effects of Manual vs Instrument-assisted Manipulation on Electromyographic Activity and Sympathetic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Nuno Filipe Pinho Nogueira, Principal Investigator, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20122018
Record Dates: First submitted 2018-11-01; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: manipulation; electromyography; sympathetic nervous system
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Double blind randomized control placebo trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Electromyographic signal and skin conductance were assessed by blinded assessors before and immediately after the intervention. The participants were not aware of their assigned group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Manual Manipulation (Experimental): A single manual manipulation was applied to C3/C4 level, on the right side.
  Interventions: Other: Manual Manipulation
- Instrument-assisted Manipulation (Active Comparator): A single instrument-assisted manipulation was applied to C3/C4 level, on the right side.
  Interventions: Other: Instrument-assisted Manipulation
- Placebo (Placebo Comparator): A placebo manipulation was applied on C3/C4 level, on the right side. The neck of th subject was placed in the pre manipulative position but no thrust was made. Then, the cervical was replaced in neutral position.
  Interventions: Other: Placebo
- Control (No Intervention): No contact was given to the subject.

INTERVENTIONS:
Other: Manual Manipulation — Subject was in supine position, and the therapist applied a manual manipulation with right side bending and left rotation of the neck.
  Arms: Manual Manipulation
Other: Instrument-assisted Manipulation — The instrument-assisted manipulation was applied using a handheld Activator IV Adjusting Instrument. Contacts were made firm enough to prevent slipping of the rubber tip but not so firm as to load the spring, in consistence with customary clinical use of the instrument. The spring was then loaded by means of the instrument's trigger mechanism, and the impulse was delivered in an anterosuperior direction, over the posterolateral aspect of the vertebra on the right lamina-pedicle junction of C3.
  Arms: Instrument-assisted Manipulation
Other: Placebo — Subject was in supine position, and the therapist placed ths subject's cervical with right side bending and left rotation but no manual manipulation was applied.
  Arms: Placebo

SUMMARY:
This study evaluates the effects of manual and instrument-assisted cervical manipulation on electromyographic activity and sympathetic nervous system. Subjects were divided in four groups, one group was submitted to a manual cervical manipulation, other group was submitted to an instrument-assisted cervical manipulation, other group was submitted to a sham manipulation and another group served as control.

DETAILED DESCRIPTION:
The manual manipulation was applied over C3/C4, as the participants were positioned in supine with the cervical spine in a neutral position. Slight ipsilateral side flexion and contralateral rotation were introduced until tension was perceived in the tissues at the contact point. A high-velocity, low-amplitude thrust manipulation was directed upward and medially in the direction of the subject's contralateral eye.

The instrument-assisted manipulation was applied using a handheld Activator IV Adjusting Instrument. Contacts were made firm enough to prevent slipping of the rubber tip but not so firm as to load the spring, in consistence with customary clinical use of the instrument. The spring was then loaded by means of the instrument's trigger mechanism, and the impulse was delivered in an anterosuperior direction, over the posterolateral aspect of the vertebra on the right lamina-pedicle junction of C3.

The sham manipulation to the right C3/C4 segment was administered using the same 'set-up' as for the manual manipulation; however, once the barrier was engaged, the head was re-positioned to neutral with no thrust applied. The control group individuals were positioned supine for the same twenty minutes as the other groups and they received no manual contact.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic individuals
* Age above 18 years.

Exclusion Criteria:

* Presence of cervical pain
* History of surgery and/neck trauma
* Osteoporosis
* Current use of anticoagulant therapy
* Presence of dizziness and/or vertigo
* Pregnancy
* Cancer
* Any other contra-indication to spinal manipulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2015-07-21 (Actual); Study Completion 2015-12-03 (Actual)

PRIMARY OUTCOMES:
Sympathetic Nervous System activity through change in skin conductance values | 10 minutes post intervention
  The effect on sympathetic nervous system was compared between manual manipulation, instrument-assisted manipulation, placebo and control. The endodermic activity amplifier Galvanic Skin Response (GSR100C) was used to collect the skin conductance values.
Change of electromyographic activity of upper trapezius after spinal manipulation | 10 minutes post intervention
  The effect on basal electromyographic activity of upper trapezius was compared between manual manipulation, instrument-assisted manipulation, placebo and control. Muscle activity was evaluated before and 10 minutes after each intervention.
Change of electromyographic activity of biceps brachii after spinal manipulation | 10 minutes post intervention
  The effect on basal electromyographic activity of biceps brachii was compared between manual manipulation, instrument-assisted manipulation, placebo and control. Muscle activity was evaluated before and 10 minutes after each intervention.